CLINICAL TRIAL: NCT04513730
Title: Development of a Positional Device Aimed at Patients With Reduced Mobility and Functional Capacity Due to Low Back Pain
Brief Title: Positional Device Aimed at Patients With Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Metodista de Piracicaba (Other)
Responsible Party: Principal Investigator, Rodrigo Santiago Barbosa Rocha, Phd, Director of Human Movement Department, Universidade Metodista de Piracicaba
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F110821
Record Dates: First submitted 2020-08-11; First posted 2020-08-14 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Rehabilitation

STUDY DESIGN:
Intervention Model Description: A device originally designed with the function of keeping the user in a comfortable position of pelvic suspension, in dorsal decubitus, with fixation in the popliteal region and ankles was built to promote lumbar traction. The device is designed in auto CAD software with 2d technical representations and 3d electronic model. It consists of a structure of PVC pipes and fittings and padded material at the support points. The structure design was based on anthropometric models according to Felisberto and Paschoarelli (2000).
  Participants belonging to both groups will receive information about the procedures performed including the objectives, risks and benefits and study protocol Participants belonging to the intervention group will be submitted to 10 pelvic suspension technique sessions using the functional prototype of the device.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pelvic suspension device (Experimental): A device will be built with the function of keeping the user in position of pelvic suspension promoting lumbar traction that will consist of a structure of pvc pipes and connections and padded material.
  Interventions: Other: Rehabilitation

INTERVENTIONS:
Other: Rehabilitation — A device originally designed with the function of keeping the user in a comfortable position of pelvic suspension, in dorsal decubitus, with fixation in the popliteal region and ankles was built to promote lumbar traction. The device is designed in autoCAD software with 2d technical representations and 3d electronic model. It consists of a structure of pipes and fittings and padded material at the support points.

SUMMARY:
The project aims to idealize a pelvic suspension device as an auxiliary physiotherapeutic resource for patients with reduced mobility and functional capacity, which should favor autonomous and independent performance in personal, social and work tasks of the target population. This is a controlled clinical trial study. The research sample will be composed of patients of both sexes, aged 21 to 65 years, diagnosed with low back pain, referred to UEAFTO/UEPA, through the SUS care network. The research participants will be evaluated by posture, active mobility and muscle strength of the spine, evaluation of pain intensity and functional capacity. A device will be built with the function of keeping the user in position of pelvic suspension promoting lumbar traction that will consist of a structure of pvc pipes and connections and padded material. Participants will be submitted to 10 sessions of use of the device, after which they will be reevaluated through the same procedures. The information collected will be analyzed through the Graphpad prism software. To compare measured values, the Shapiro-Wilk test will be used for normality distribution. Student's t-tests will be used for the treatment of variables with normal distribution, and Fisher's and Mann-Whitney's exact tests for variables without normal distribution. It is expected to collaborate in the social integration, labor and quality of life of people affected by low back pain, as well as to promote the development of low-cost technologies in the routine of Physiotherapy and public health in the State of Pará.

ELIGIBILITY:
Inclusion Criteria:

* patients with low back pain

Exclusion Criteria:

* patients with a history of vertebral surgery
* patients with spinal tumors
* patients with intervertebral disc infections
* patients with vertebral fractures
* patients with severe osteoporosis
* patients with ankylosing processes of the spine
* patients with heart diseases

Ages: 25 Years to 61 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2020-08-11 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Lumbar dynamometry | post treatment in 3 days
  The dynamometer is an instrument used to assess muscle strength in individuals with normal health status and/or in the process of rehabilitation (EICHINGER et al., 2015). The lumbar dynamometer has the function of measuring the isometric strength of the extensor musculature of the Lumbar spine. The participant is positioned standing on the platform of the equipment with total extension of knees, trunk in flexion with about 120º and the head accompanies the extension of the trunk, the hands hold the dynamometer bar positioned previously. For learning, the participant performs two to three subm maxima contractions. Then, the maximum contraction is requested in 3 attempts with one minute of rest
Photogrammetric goniometry | post treatment in 3 days
  Active mobility of the lumbar spine will be evaluated by means of photogrammetry with the same instruments of postural assessment. The flexion, extension, and lateral flexion movements on the right and left will be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade do Estado do Pará, Belém, Pará, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Mataran-Penarrocha GA, Lara Palomo IC, Antequera Soler E, Gil-Martinez E, Fernandez-Sanchez M, Aguilar-Ferrandiz ME, Castro-Sanchez AM. Comparison of efficacy of a supervised versus non-supervised physical therapy exercise program on the pain, functionality and quality of life of patients with non-specific chronic low-back pain: a randomized controlled trial. Clin Rehabil. 2020 Jul;34(7):948-959. doi: 10.1177/0269215520927076. Epub 2020 Jun 10. PMID 32517498
- [Result] Hayden JA, Wilson MN, Stewart S, Cartwright JL, Smith AO, Riley RD, van Tulder M, Bendix T, Cecchi F, Costa LOP, Dufour N, Ferreira ML, Foster NE, Gudavalli MR, Hartvigsen J, Helmhout P, Kool J, Koumantakis GA, Kovacs FM, Kuukkanen T, Long A, Macedo LG, Machado LAC, Maher CG, Mehling W, Morone G, Peterson T, Rasmussen-Barr E, Ryan CG, Sjogren T, Smeets R, Staal JB, Unsgaard-Tondel M, Wajswelner H, Yeung EW; Chronic Low Back Pain IPD Meta-Analysis Group. Exercise treatment effect modifiers in persistent low back pain: an individual participant data meta-analysis of 3514 participants from 27 randomised controlled trials. Br J Sports Med. 2020 Nov;54(21):1277-1278. doi: 10.1136/bjsports-2019-101205. Epub 2019 Nov 28. PMID 31780447
- [Result] Calatayud J, Escriche-Escuder A, Cruz-Montecinos C, Andersen LL, Perez-Alenda S, Aiguade R, Casana J. Tolerability and Muscle Activity of Core Muscle Exercises in Chronic Low-back Pain. Int J Environ Res Public Health. 2019 Sep 20;16(19):3509. doi: 10.3390/ijerph16193509. PMID 31547140
- [Result] Suso-Ribera C, Camacho-Guerrero L, Osma J, Suso-Vergara S, Gallardo-Pujol D. A Reduction in Pain Intensity Is More Strongly Associated With Improved Physical Functioning in Frustration Tolerant Individuals: A Longitudinal Moderation Study in Chronic Pain Patients. Front Psychol. 2019 Apr 26;10:907. doi: 10.3389/fpsyg.2019.00907. eCollection 2019. PMID 31133917
- [Result] Arguisuelas MD, Lison JF, Domenech-Fernandez J, Martinez-Hurtado I, Salvador Coloma P, Sanchez-Zuriaga D. Effects of myofascial release in erector spinae myoelectric activity and lumbar spine kinematics in non-specific chronic low back pain: Randomized controlled trial. Clin Biomech (Bristol). 2019 Mar;63:27-33. doi: 10.1016/j.clinbiomech.2019.02.009. Epub 2019 Feb 14. PMID 30784788